CLINICAL TRIAL: NCT06237478
Title: Effects of Glycopyrrolate on Heart Rate and Heart Rate Variability in Patients With Different Basic Heart Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20240123
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Glycopyrrolate
Keywords: Glycopyrrolate; Heart rate; Heart rate variability; Autonomic nervous system
MeSH Terms: interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): The HR at 10 minutes after the start of surgery was considered as the baseline HR. Patients were divided into two groups based on their baseline HR: Group L: Baseline HR 40-60 beats/min.
  Interventions: Drug: Glycopyrrolate
- Group H (Experimental): The HR at 10 minutes after the start of surgery was considered as the baseline HR. Patients were divided into two groups based on their baseline HR: Group H: Baseline HR 60-100 beats/min.
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Glycopyrrolate — At the timepoint of 10 min after operation beginning (T1), the basic HR, MAP and the HRV frequency indexes were recorded. Then glycopyrrolate 0.006 mg/kg was injected intravenously in Group L.
  Arms: Group L
Drug: Glycopyrrolate — At the timepoint of 10 min after operation beginning (T1), the basic HR, MAP and the HRV frequency indexes were recorded. Then glycopyrrolate 0.006 mg/kg was injected intravenously in Group H.
  Arms: Group H

SUMMARY:
Glycopyrrolate is an anticholinergic medication commonly used in respiratory medicine for treating chronic obstructive pulmonary disease (COPD), bronchial asthma, and other conditions . In the perioperative period, it is often administered before anesthesia to reduce secretions in the salivary glands, bronchi, and pharynx . It is used during the recovery period to counteract the muscarinic effects of anticholinesterase inhibitors and can also be employed to prevent/treat vagal reflexes and related arrhythmias induced by surgery or medications .

Heart rate (HR) is influenced by both the sympathetic and parasympathetic nervous systems. The baseline HR of different patients may vary due to differing levels of sympathetic and parasympathetic nerve activity within the body. It remains unclear whether patients with different baseline HRs exhibit varying degrees of HR elevation after the administration of glycopyrrolate(i.e.,the parasympathetic activity in vivo is antagonized). The primary aim of this study is to explore the impact of glycopyrrolate administration on HR in patients with different baseline HRs. The secondary objective is to investigate the effects of glycopyrrolate on heart rate variability (HRV) in patients with different baseline HR.

ELIGIBILITY:
Inclusion Criteria:

* 1.Weight not restricted; 2.American Society of Anesthesiologists (ASA) status I or II; 3.The operative time≥1 h; 4.Undergoing orthopedic or urological surgery.

Exclusion Criteria:

* 1.allergy to glycopyrrolate; 2.laparoscopic surgery; 3.liver or kidney dysfunction; 4.pre-existing abnormal electrocardiogram such as bradycardia; 5.concomitant glaucoma; 6.patients refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The maximum increase of HR | before induction of general anesthesia; 10 min after operation beginning; 30 min after glycopyrrolate injection
  Calculation of the maximum increase of HR (∆HR): The increase in heart rate (HR) at 30 minutes after the administration of glycopyrrolate (T2) compared to 10 minutes after the start of surgery (T1) was calculated as the maximum increase of HR.
the maximum increase ratio of HR | before induction of general anesthesia; 10 min after operation beginning; 30 min after glycopyrrolate injection
  The maximum increase ratio of HR =∆HR/[HR at T1]) .

SECONDARY OUTCOMES:
HRV frequency indexes | before induction of general anesthesia; 10 min after operation beginning; 30 min after glycopyrrolate injection
  HRV frequency indexes included Low frequency power (LF, 0.04-0.15 Hz), High frequency power (HF, 0.15-0.4 Hz) and LF/HF.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China